CLINICAL TRIAL: NCT00220012
Title: Effect of Folate on Colonic and Blood Cells
Brief Title: Effect of Folate on Colon and Blood Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PHO-0514; N01-CN-35111
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Subjects Will Have a Pre-cancerous Colorectal Polyp; Family Member Has History of Colorectal Adenoma of Adenocarcinoma
MeSH Terms: interventions — Dietary Supplements

INTERVENTIONS:
Procedure: Folate depletion and supplementation

SUMMARY:
This study looks at the effect of folate supplementation and depletion on the blood cells and the colorectal cells. To examine the effect of these changes, blood samples and colorectal biopsy samples are collected. The genetic material (RNA and DNA) is examined to see what changes occur during the depletion and supplementation of folate. The hypothesis is that folate may help prevent colon cancer

DETAILED DESCRIPTION:
Folate Depletion Arm and Supplementation Arm:

The folate depletion study requires an 8-week run-in period. During this run-in period, all participants will eat an average folate diet with no high folate containing foods. There are two screening visits during this period where initial blood-work is done and participants undergo nutritional consultation. Following the 8-week run-in period, subjects in the folate depletion arm will be hospitalized for approximately 3 months at the Rockefeller University Hospital. You may leave the hospital during the day, but are required to return each evening. During this entire time, subjects are given a low folate diet. During the last month of the study, folate supplements are given to replace folate in the body. A follow-up visit is required approximately 1 month after the study period. Blood will be drawn every two weeks. Four sigmoidoscopies will be taken at approximately monthly intervals. A male is required to use an effective form of birth control throughout his participation in the study and for two months after the study ends.

The folate supplementation study requires an 8-week run-in period. During this run-in period, all participants will eat an average folate diet with no high folate containing foods. There are two screening visits during this period where initial blood-work is done and participants undergo nutritional consultation. Following the 8-week run-in period, subjects in the folate supplementation arm will be given a folate supplement for 8 weeks. During this entire time, subjects will continue to eat an average folate diet with no high folate containing foods. Blood samples and colorectal mucosa samples obtained during a sigmoidoscopy will be taken 3 times at 4 week intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Men or post-menopausal women ages 40 to 72 years old that have a personal history of colorectal adenomatous polyps and/or have a family history of colorectal cancer or polyps will be included. Women have to be ≥2 years post-menopause (2 years after the last menstrual period).
2. Ambulatory and in good health. -

Exclusion Criteria:

* 1. Personal history of cancer other than non-melanoma skin cancer.

  2. History of hereditary non-polyposis colon cancer or more that one first degree family member with colorectal or endometrial cancers.

  3. Diseases of the bowel such as intestinal malabsorption or inflammatory bowel disease

  4. Surgery to the stomach or colon not including removal of the appendix or surgery to the esophagus (food tube)

  5. Any excessive bleeding or clotting disorder or if you are taking blood thinners.

  6. Abnormalities of or conditions predisposing you to abnormalities of, folate metabolism.

  7. Untreated hyperthyroidism (increase in thyroid function) or insulin-requiring diabetes mellitus

  8. Daily alcohol intake greater than 2 ½ shot glasses of whisky or three -8 ounce glasses of beer or wine.

  9. No regular dosing of 660 mg of aspirin per day or more than 660 mg per day

This is equal to or more than two tablets of 325 mg. of regular strength aspirin; or equal to or more than one tablet of 500 mg. extra-strength aspirin. You must not have regularly taken dosages of nonsteroidal anti-inflammatory agents (NSAID's) within the last 3 months. One example of an NSAID is ibuprofen.

If you have been taking aspirin for heart or blood vessel protection regularly for at least one month before your first screening visit, you will remain on that same amount of medicine throughout the study and is allowed as follows:

* Aspirin 1 to 2 regular aspirin tablets (325 mg per tablet) per day, or
* Baby aspirin per day (81mg tablet).

  10. A blood level (plasma) Vitamin B12 level less than 250pg/mL or a folate level greater than 20 ng/ml

  11. A blood (plasma) homocysteine level equal to or greater than 17 μmol/L

  12. Taking a medication called, sterol-binding resins, such as cholestyramine (Questran ®), which is for the treatment of high blood cholesterol.

  13. Taking other investigational medications or multiple other medications that might, in the opinion of the investigator, alter cell production in your rectum; folate metabolism, or kidney or liver metabolism.

  14. Any serious illness that would be anticipated to limit life expectancy to less than 6 months

  15. Sustained elevated blood pressure greater than 150/95 mm Hg for three consecutive readings.

  16. Clinically significant liver disease as evidenced by blood levels of alanine amniotransferase or aspartate amniotransferase, greater than two times the upper limits of the normal range, unexplained elevated alkaline phosphatase, or kidney disease with blood creatinine level greater than 2.0 mg/dL.

  17. HIV positive test results.

  18. Currently taking any of the following:
* Weight control medications.
* Folic acid containing medications greater than 400 micrograms per day.
* Hormone replacement therapies or oral, transplanted, and injected contraceptives.
* Thyroid hormone replacement medications

  o These will be only allowed if you have been stable on thyroid medication (euthyroid) for three months.
* Medication interfering with the folic acid metabolic effects such as methotrexate (includes Folex® and Trexall® and others), antiepileptic drugs such as phenytoin (Dilantin®), phenobarbital, primidone or sulfonamides (includes some antimicrobial agents) and folinic acid derivatives (Leucovorin®).
* Lipid-lowering medications (with the following exceptions)

If you have been taking the following lipid lowering medication of the class called "statins" regularly for at least one month before your first screening visit, you will remain on the same amount of medicine throughout the study.

* Atorvastatin (Lipitor©) 10 or 20 mg/day
* Fluvastatin (Lescol©) 20 mg or 40 mg/day
* Lovastatin (Levacor©) 10 or 20 mg/day
* Pravastatin (Pravachol©) 10 or 20 mg/day
* Simivastatin (Zocor©) 5 or 10 mg/day

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-06; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Measurements of established folate-related endpoints in DNA from blood mononuclear cells and rectal cells:
Luracil incorporation in blood mononuclear cells
Strand breaks in the coding region of p53 in blood cells and rectal biopsy cells
DNA methylation (overall, p53, coding, p16 promotor. MLH1 promotor) in blood cells and rectal biopsy cells

SECONDARY OUTCOMES:
Measurements of differential gene expression in colonic and blood cells by microarray analysis, further defining folate's action in modifying cell cycle activity, cell maturation, signal transduction and oncogene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Holt, MD, Principal Investigator — Rockefeller University and Strang Cancer Institute
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Derived] Protiva P, Mason JB, Liu Z, Hopkins ME, Nelson C, Marshall JR, Lambrecht RW, Pendyala S, Kopelovich L, Kim M, Kleinstein SH, Laird PW, Lipkin M, Holt PR. Altered folate availability modifies the molecular environment of the human colorectum: implications for colorectal carcinogenesis. Cancer Prev Res (Phila). 2011 Apr;4(4):530-43. doi: 10.1158/1940-6207.CAPR-10-0143. Epub 2011 Feb 14. PMID 21321062
- See also: Related Info — http://www.rucares.org